CLINICAL TRIAL: NCT06424145
Title: A Single-center, Randomized and Controlled Clinical Research Projects
Brief Title: Effect of Local Anesthesia Position of Lidocaine Injection on the Success Rate of Radial Artery Puncture Tube
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ting Xu (Other)
Responsible Party: Sponsor-Investigator, Ting Xu, Chief physician, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19981228
Record Dates: First submitted 2024-05-01; First posted 2024-05-21 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Radial Artery Injury
Keywords: Puncture site of radial artery; Lidocaine injection; Success ratio; Invasive blood pressure measurement; Radial artery puncture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superior group of radial artery (Experimental): Injection of 1% lidocaine 1 ml above the artery
  Interventions: Diagnostic Test: Superior radial artery
- Right radial artery group (Experimental): Injection of 1% lidocaine 1 ml to the right side of the artery
  Interventions: Diagnostic Test: Right side of radial artery

INTERVENTIONS:
Diagnostic Test: Superior radial artery — Upper radial artery, 1 ml of lidocaine
  Arms: Superior group of radial artery
Diagnostic Test: Right side of radial artery — Right side of the radial artery,1ml of lidocaine
  Arms: Right radial artery group

SUMMARY:
Objective: To investigate the effect of lidocaine injection location on the success rate of ultrasound-guided radial artery catheterization in a single-center, randomized, controlled clinical trial.

DETAILED DESCRIPTION:
Group A was randomly divided into two groups: 1% lidocaine 1 ml was injected above the artery during local anesthesia before arterial catheterization; Group B: 1ml of 1% lidocaine was injected into the right side of the artery. The proportion of subjects according to the number of PO was similar in all groups. After the screening, the scientific research personnel of each testing center will log in the random system, fill in the screening information, obtain the random number information, and distribute the corresponding scientific research drugs according to the random number. The total number of drugs is imported into the centralized random grouping system by generating random number by SAS software. The study was conducted by an evaluation researcher and a medication management researcher. Throughout the experiment, not only the subjects turned a blind eye, but also the evaluators turned a blind eye. This study set up evaluation investigators and administrative investigators. Administrative researchers were only involved in the randomization, allocation, and delivery process. Other procedures, including informed consent, screening, efficacy index and safety evaluation, and planned visits, were completed by the evaluation investigators.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Class I-III, patients aged 18-80 years
2. Planned surgery with radial artery catheterization
3. Allen test negative
4. Sign the informed consent form and voluntarily participate in this trial

Exclusion Criteria:

1. Inflamed skin at puncture site
2. Extremely nervous and unable to cooperate
3. Ultrasonographic assessment of aberrant radial artery
4. Significant abnormalities in coagulation function (PT prolongation exceeding the upper limit of normal for 3 s or APTT prolongation exceeding the upper limit of normal for 10 s)
5. The patient had undergone radial artery catheterization in the same arm in the past week
6. History of hypersensitivity to local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Success ratio of first radial artery puncture | Day 1
  What is the probability of success the first time?

SECONDARY OUTCOMES:
Before and after lidocaine local anesthesia, the radial artery longest diameter and shortest diameter, circumference, cross-sectional area and depth changes | Day 1
  In millimeters, Increase or decrease

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan provincial Peopel'Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No